CLINICAL TRIAL: NCT01766011
Title: Evaluation of a Standard Preterm Infant Formula Fed to Preterm Infants in the Hospital
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AL01
Record Dates: First submitted 2013-01-08; First posted 2013-01-11 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Pre-term Infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- study pre-term formula (Experimental): Pre-term formula with a modified stabilizer system in 2 oz. ready to feed plastic bottles
  Interventions: Other: study pre-term formula

INTERVENTIONS:
Other: study pre-term formula — 24 kcal/fl oz pre-term formula for in-hospital use
  Other Names: Similac Special Care

SUMMARY:
The purpose of this study is to assess overall growth of preterm infants fed a reformulated preterm infant formula during hospitalization. All study products meet levels of nutrients for the infant population as specified in the Infant Formula Act and all subsequent amendments.

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible for study participation will satisfy the following criteria:

  * Birth weight between 1000g -1800g
  * Less than or equal to 34 weeks and 0 days gestational age at birth
  * Appropriate for gestational age (AGA)
  * Singleton or twin births
  * Infant is 21 days of age or less

Exclusion Criteria:

* Infants with the following conditions prior to and/or at the time of study product initiation are not eligible for entry into the study:

  * Expected to be transferred to another facility within 14 days
  * Serious congenital abnormalities that may affect growth and development
  * Intubated for ventilation at the time of study product initiation
  * Grade III or IV periventricular/intraventricular hemorrhage (PVH/IVH)
  * Maternal incapacity, maternal drug or alcohol abuse during pregnancy or current abuse, or maternal treatment consistent with human immunodeficiency virus therapy
  * Infant has a history of major surgery
  * Asphyxia defined as progressive hypoxemia and hypercapnia with significant metabolic acidemia
  * Confirmed necrotizing enterocolitis or confirmed sepsis
  * Current use or planned use of probiotics
  * Participation in another study that has not been approved

Max Age: 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2012-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Weight gain per day | Study Day (SDAY) 1 to SDAY 29, or hospital discharge, whichever comes first
  weight gain per day (g/kg/d)

SECONDARY OUTCOMES:
Length | Study Day (SDAY) 1 to SDAY 29, or hospital discharge, whichever comes first
  Growth, change in length
Daily Stool Questionnaire | Study Day (SDAY) 1 to SDAY 29, or hospital discharge, whichever comes first
  Gastro-intestinal Tolerance; Presence of bloody, watery, hard or black stools will be captured.
Serum Calcium | SDAY 1, 15, and 29 or hospital discharge (whichever comes first)
  Blood biochemistries
Head circumference | Study Day (SDAY) 1 to SDAY 29, or hospital discharge, whichever comes first
  Growth, change in head circumference
Daily Feeding Questionnaire | Study Day (SDAY) 1 to SDAY 29, or hospital discharge, whichever comes first
  Gastro-Intestinal Tolerance; Cause for withholding feedings will be captured.
Any periods of nil per os (NPO) | Study Day (SDAY) 1 to SDAY 29, or hospital discharge, whichever comes first
  Gastro-Intestinal Tolerance
Phosphorus | SDAY 1, 15, and 29 or hospital discharge (whichever comes first)
  Blood biochemistries
Alkaline Phosphatase | SDAY 1, 15, and 29 or hospital discharge (whichever comes first)
  Blood biochemistries

CONTACTS AND LOCATIONS:
Overall Officials: Bridget Barrett Reis, PhD, RD, LD, Study Chair — Abbott Nutrition
Locations (7):
- United States (7):
  - University of South Alabama - Children's and Women's Hospital, Mobile, Alabama
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Wesley Medical Center, Wichita, Kansas
  - Maria Children's Hospital Westchester Medical Center, Valhalla, New York
  - MetroHealth Medical Center, Cleveland, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Wheaton Franciscan Healthcare-St. Joseph, Milwaukee, Wisconsin